CLINICAL TRIAL: NCT06936488
Title: A Prospective, Single Arm, Open Label, Phase II Clinical Study on the Efficacy and Safety of Ivonescimab (AK112) Combined With TAS-102 in the Treatment of Refractory MSS/pMMR Advanced Colorectal Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HACRC-01
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-12

CONDITIONS: MSS/pMMR Type Metastatic Colorectal Adenocarcinoma Patients
Keywords: intestinal cancer，Ivonescimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab (Experimental)
  Interventions: Drug: Ivonescimab,TAS-102

INTERVENTIONS:
Drug: Ivonescimab,TAS-102 — Ivonescimab,20mg/kg,i.v.,D1,Q3w TAS-102,35mg/m2,bid,D1-5,Q2W

SUMMARY:
A Prospective, Single Arm, Open Label, Phase II Clinical Study on the Efficacy and Safety of Ivonescimab (AK112) Combined With TAS-102 in the Treatment of Refractory MSS/pMMR Advanced Colorectal Cancer

Main purpose:

Evaluate the efficacy and safety of the combination therapy of Ivonescimab (AK112) and TAS-102 in the treatment of refractory MSS/pMMR advanced colorectal cancer

Exploratory purpose:

Evaluation of the relationship between immune markers, patient efficacy, and prognosis in the treatment of refractory MSS/pMMR advanced colorectal cancer with the combination of Ivonescimab (AK112) and TAS-102 Study endpoint

Primary endpoint:

Researchers evaluated the PFS rate at 18 weeks based on RECIST v1.1.

Secondary endpoint:

ORR, DCR, PFS, and OS evaluated based on RECIST v1.1. The incidence and severity of adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old and above but 75 years old and below, regardless of gender;
2. Previously received at least two standard chemotherapy regimens for advanced colorectal cancer and demonstrated disease progression or intolerance to the last regimen.

   Patients who have received adjuvant/neoadjuvant chemotherapy and experience recurrence during or within 6 months after completion of adjuvant/neoadjuvant chemotherapy can be considered as a chemotherapy regimen for advanced disease;
3. There are sufficient tissue specimens that have been tested as pMMR (immunohistochemistry) or MSS (PCR or NGS)
4. Have at least one measurable lesion (RECIST v1.1);
5. ECOG PS score is 0 or 1;
6. Expected survival exceeds 3 months;
7. The main organ functions are normal, which meets the following criteria:

   Absolute neutrophil count ≥ 1.5 x 10 ^ 9/L Hemoglobin ≥ 9 g/dL Platelet count ≥ 100 x 10 ^ 9/L Creatinine clearance rate ≥ 50 mL/min, evaluated using the Cockcroft&Gault formula Serum total bilirubin<1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) ≤ 2.5 x ULN (unless liver metastasis leads to abnormal liver function, aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 5 x ULN) All patients have normal coagulation function. For patients receiving anticoagulant therapy (excluding platelet anticoagulants), it should be confirmed that the INR has reached a sufficient therapeutic level.
8. The subjects voluntarily joined this study and signed informed consent forms, demonstrating good compliance and cooperation with follow-up;
9. Women with fertility: must agree to use reliable methods of contraception for at least 180 days from the signing of the informed consent form until the last administration of the study drug. And the serum HCG test must be negative within 7 days before starting the study treatment; And it must be non lactating. If a female patient has already menstruated, has not yet reached postmenopausal status (continuous absence of menstruation for ≥ 12 months, no other reasons found besides menopause), and has not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), it is considered that the patient has fertility;
10. For male patients whose partners are women with fertility, they must agree to use reliable methods of contraception for at least 180 days from the signing of the informed consent form until the last administration of the study drug. Male patients must also agree not to donate sperm during the same time period.

Exclusion Criteria:

1. Previously received TAS-102 treatment.
2. Previously received immunotherapy, including immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, anti-CD47 antibodies, anti-SIRP α antibodies, anti-LAG-3 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immunotherapy, and any other treatment targeting the immune mechanism of tumor.
3. Severe wounds that do not heal, ulcers that do not heal, or fractures that do not heal.
4. Known coagulation disorders and bleeding disorders that increase the risk of bleeding.
5. Researchers believe that patients are unlikely to comply with oral medication treatment plans or study requirements for scheduled evaluations.
6. Pregnant, lactating women or those who may become pregnant during the study period.
7. Symptomatic central nervous system metastasis with unstable nervous system or the need to increase steroid dosage to control central nervous system diseases.
8. Suffering from severe or uncontrolled active acute or chronic infections.
9. Suffering from interstitial lung disease and/or pneumonia, or pulmonary arterial hypertension.

Researchers believe that uncontrolled arterial hypertension or uncontrolled or symptomatic arrhythmia.

11. Study whether there have been deep arterial thromboembolic events, including cerebrovascular accidents or myocardial infarction, within 6 months prior to the start of the first treatment. Study the occurrence of deep vein thromboembolism events within 4 weeks prior to the first treatment.

12. Severe/unstable angina, symptomatic congestive heart failure, New York Heart Association (NYHA) class III or IV.

13. Other malignant tumors, including those that have received curative treatment and have a remission period of less than 5 years during screening. Patients with cervical carcinoma in situ and basal cell carcinoma who can be cured with appropriate treatment are exempt from this minimum required remission period.

Receive systemic immunosuppressive therapy (excluding prophylactic or long-term low-dose steroids [≤ 20 mg/day prednisone equivalent]).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS rate at 18 weeks | At the end of Cycle 6 (each cycle is 28 days)
  The progression free survival rate (PFS) at 18 weeks refers to the proportion of patients who have experienced objective deterioration or progression (including death) of the disease for the first time since the start of treatment, and whose survival time has reached or exceeded 18 weeks

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of Cycle 6 (each cycle is 28 days)
  The ORR is defined as the proportion of patients with a response of CR or PR
Overall survival (OS) | From date of randomization to death from any cause, assessed up to 2 years
  From the date of randomization until the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University#Huai'an First People's Hospital#, Huai'an, Jiangsu, China